CLINICAL TRIAL: NCT00059813
Title: A Phase II Trial of G3139 (Genasense) Anti-Bcl-2 Antisense Oligonucleotide Plus Alpha-Interferon in Metastatic Renal Cancer
Brief Title: Oblimersen and Interferon Alfa in Treating Patients With Metastatic Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02828; NCI-2012-02828 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-42 (Other: City of Hope); 5828 (Other: CTEP); N01CM17101 (NIH)
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Recurrent Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Interferon-alpha; Interferon Alfa-n3; Introns; Interferon alpha-2; oblimersen

ARMS (1):
- Treatment (recombinant interferon alfa, oblimersen sodium) (Experimental): Patients receive oblimersen IV continuously on days 1-7 and interferon alfa subcutaneously on days 4, 6, 8, 10, and 12 of course 1 and on days 1, 3, 5, 8, 10, and 12 of all subsequent courses. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. Patients achieving a CR receive an additional 2 courses past CR.
  Interventions: Biological: recombinant interferon alfa; Biological: oblimersen sodium; Other: pharmacological study

INTERVENTIONS:
Biological: recombinant interferon alfa — Given SC
  Other Names: Alferon N; alpha interferon; IFN-A; Intron A; Roferon-A
Biological: oblimersen sodium — Given IV
  Other Names: augmerosen; G3139; G3139 bcl-2 antisense oligodeoxynucleotide; Genasense
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase II trial to study the effectiveness of combining oblimersen with interferon alfa in treating patients who have metastatic renal cell (kidney) cancer. Interferon alfa may interfere with the growth of tumor cells. Oblimersen may increase the effectiveness of interferon alfa by making tumor cells more sensitive to the drug.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the objective response rate of metastatic renal cancer to the combination of G3139 plus α-Interferon (α-IFN).

SECONDARY OBJECTIVES:

I. To further assess the clinical toxicity of this combination. II. To evaluate the impact of G3139 plus α-IFN on molecular targets involved in the regulation of apoptosis in tumor cells and lymphocytes.

III. To evaluate the pharmacokinetics of G3139 when given with α-IFN at this dose and schedule.

IV. To evaluate the potential toxicity of this combination on cells of the immune system.

OUTLINE: This is a multicenter study.

Patients receive oblimersen IV continuously on days 1-7 and interferon alfa subcutaneously on days 4, 6, 8, 10, and 12 of course 1 and on days 1, 3, 5, 8, 10, and 12 of all subsequent courses. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete remission (CR) receive an additional 2 courses past CR.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 21-41 patients will be accrued for this study within 20-24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, measurable metastatic renal cell cancer; if a nephrectomy was performed in the setting of metastatic disease, post-nephrectomy progression of metastases must be documented
* Performance status 0-2 (SWOG), life expectancy > 3 months
* Prior radiation must have been completed > 4 weeks before enrollment, with measurable disease outside of the radiation port
* WBC > 3500/μl
* Absolute neutrophil count > 1500/μl
* Platelets > 100,000/μl
* Transaminases < 2 x institutional upper limit of normal
* Serum bilirubin < 1.5 x institutional upper limit of normal (if Gilbert's, up to 2 x upper limit)
* Serum alkaline phosphatase < 2.5 x institutional upper limit of normal
* Patients with hepatic metastases may have 50% higher levels of all the above-listed parameters
* Serum creatinine < 1.5 x institutional upper limit of normal
* Patients with active or recently-treated autoimmune disease are excluded, as are patients currently receiving or expected to require corticosteroid therapy
* Prior malignancy is limited to adequately treated non-melanoma skin cancer, cervical carcinoma-in-situ, or any other malignancy for which the patient has been disease-free for at least 5 years
* Because the effects of G3139 on the unborn fetus or newborn infant are unknown, pregnant or lactating women are excluded, and patients with reproductive potential must agree to use a medically-acceptable form of birth control
* Patients must have fully recovered from the effects of any prior surgery or medical illness such as infection; those with psychosocial problems that might compromise safety or protocol compliance are excluded
* Central venous access is required
* Patients may have received up to two prior biological therapy regimens, excluding exposure to either of the therapy agents and patients may have had no more than one prior chemotherapy regimen; full recovery from all toxicities must have occurred; for high-dose IL-2, at least 8 weeks must have elapsed since prior treatment
* Written, voluntary informed consent
* Previous chemotherapy must have been completed at least 3 weeks before treatment under this protocol can be initiated
* Patients with a history of brain metastases, or who are currently being treated, or have untreated brain metastases, are not eligible; Note: if patient received steroid therapy, at least three weeks must have elapsed prior to entry on this protocol
* Patients must have normal baseline PT/PTT; Note: For those patients taking low dose coumadin (e.g., as prophylaxis for a venous access device) and INR of up to 1.5 is allowed

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2003-08; Primary Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Objective response rate based on the Response Evaluation Criteria In Solid Tumors (RECIST) | Start of the treatment until disease progression/recurrence, assessed up to 5 years
  Confidence intervals for the response rate will be established by calculating exact 95% confidence limits for a binomial parameter.

SECONDARY OUTCOMES:
Overall survival | Time from first day of treatment to time of death due to any cause, assessed up to 5 years
  Estimated using the product-limit method of Kaplan and Meier.
Progression free survival | Time from first day of treatment to the first observation of disease progression or death due to any cause, assessed up to 5 years
  Estimated using the product-limit method of Kaplan and Meier.
Time to progression | Time from first day of treatment to the first observation of disease progression or death due to disease, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kim Margolin, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States